CLINICAL TRIAL: NCT02245529
Title: Secotex ®: Prescription Event Monitoring in Patients With Benign Prostatic Hyperplasia (BPH)
Brief Title: Safety Profile of Secotex ® in Patients With Benign Prostatic Hyperplasia
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 527.64
Record Dates: First submitted 2014-09-18; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tamsulosin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with benign prostatic hyperplasia (BPH)
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: Tamsulosin
  Other Names: Secotex ®

SUMMARY:
The Objective of this study is to conduct a Prescription Event Monitoring (PEM) involving patients treated with Secotex® (Tamsulosin) in "real life" settings. The aim of a PEM is to monitor the safety profile of Secotex® in a cohort of patients with Benign Prostatic Hyperplasia as used in general practice

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age with a diagnosis of symptomatic Benign Prostatic Hyperplasia (BPH) and/or that, according to the Physician, their symptoms require medical treatment to improve their quality of life. The patients could be naïve to treatment or could be on treatment with other drugs but have not responded adequately to treatment. This study is non-interventional, so the decision to treat must be based on the best standard accepted clinical practice, and according to Secotex® prescribing information

Exclusion Criteria:

* Patients with known hypersensitivity to Tamsulosin, or any other component of the product
* Patients with a history of orthostatic hypotension or severe liver failure

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of symptomatic Benign Prostatic Hyperplasia (BPH) who require medical treatment to improve their quality of life
Sampling Method: Non-Probability Sample
Enrollment: 982 (Actual)
Dates: Start 2005-03; Primary Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to 6 months